CLINICAL TRIAL: NCT01021644
Title: Effects of Standardized Aerobic Exercise-Training on Neurocognitive and Neurodegeneration
Brief Title: Genes, Exercise, Memory and Neurodegeneration
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Howard University (Other)
Responsible Party: Principal Investigator, Thomas Obisesan, Professor of Medicine, Howard University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IA0172; 1R01AG031517-01A209; 1R01AG031517-01 (NIH)
Record Dates: First submitted 2009-11-25; First posted 2009-11-30 (Estimated); Last update posted 2014-02-14 (Estimated); Status verified 2014-02

CONDITIONS: Alzheimer's Disease
Keywords: APOE; Apolipoprotein E; Cognition Disorders; Neurocognition
MeSH Terms: conditions — Alzheimer Disease; Cognition Disorders | interventions — Plyometric Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- aerobic exercise-training (Experimental)
  Interventions: Behavioral: aerobic exercise-training
- stretch exercise (Active Comparator)
  Interventions: Behavioral: stretch exercise

INTERVENTIONS:
Behavioral: aerobic exercise-training — 3 times per week for 6 months
  Arms: aerobic exercise-training
Behavioral: stretch exercise — 3 times per week for 6 months
  Arms: stretch exercise

SUMMARY:
The primary purpose of this pilot study is to determine whether African Americans with mild Alzheimer's disease (AD) can be enrolled and retained in a 6-month aerobic exercise-training study.

DETAILED DESCRIPTION:
This study will examine the effects of aerobic exercise-training on neurocognitive function, and on cerebral glucose homeostasis. It is yet to be determined whether African Americans with mild AD can be recruited into such a study, nor has the relationship of fitness adaptation to neurocognitive function been systematically examined in this population. In addition to the goal of assessing the intervention effects, the study will evaluate the differential relationships of APOE to aerobic fitness-induced changes in neurocognition. The long-term goal is to explore the mechanism by which fitness adaptation exerts an effect on neurocognition, notably, low levels of high-density lipoprotein cholesterol (HDL-C), elevated inflammation (C-reactive protein (CRP) and interleukins (IL-1A)), deranged glucose homeostasis, hypertension and endothelia dysfunction are precursors of arteriolosclerosis, decreased cerebral perfusion and oxygen deprivation, all of which may increase AD risk. Because many of these putative AD risk factors are susceptible to lifestyle alterations, the study will also assess their roles in aerobic fitness-related improvements in cognitive function and reduction in AD risk.

ELIGIBILITY:
Inclusion Criteria:

* Age over 60 years
* Ability to exercise vigorously without harm
* Mild AD
* Study partner
* In good general health
* Willing to exercise for 6 months
* Body Mass Index (BMI) less than 37
* Women participants must be postmenopausal for at least 2 years, and maintain current hormone replacement therapy status and allowed medication usage for the duration of the study

Exclusion Criteria:

* MMSE score below 20
* TG (Triglyceride) greater than 400 mg/dl
* LDL-C levels greater than 95% or HDL-C levels less than 10% of age and sex-adjusted norms

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2009-10; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
AD Assessment Scale-Cognitive (ADAS-COG) | baseline, 3 and 6 months

SECONDARY OUTCOMES:
Mini-Mental State Exam (MMSE) | baseline, 3 and 6 months
CDR (Clinical Dementia Rating) Scale | baseline, 3 and 6 months
Logical Memory Test (Delayed Paragraph Recall) | baseline and 6 months
Visuospatial and Visuographic: Clock Drawing Test | baseline and 6 months
American National Adult Reading Test (ANART) | baseline and 6 months
Neuropsychiatric Inventory Q (NPIQ) | baseline and 6 months
Geriatric Depression Scale | baseline and 6 months
Activities of Daily Living (ADCS-ADL) | baseline and 6 months
PET imaging to measure cerebral glucose homeostasis/metabolism | baseline and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Thomas O. Obisesan, MD, MPH, Principal Investigator — Howard University
Locations (2):
- United States (2):
  - Howard University General Clinical Research Center (GCRC), Washington D.C., District of Columbia
  - Temple University Exercise Physiology Laboratory, Philadelphia, Pennsylvania

REFERENCES:
- [Background] Lautenschlager NT, Cox KL, Flicker L, Foster JK, van Bockxmeer FM, Xiao J, Greenop KR, Almeida OP. Effect of physical activity on cognitive function in older adults at risk for Alzheimer disease: a randomized trial. JAMA. 2008 Sep 3;300(9):1027-37. doi: 10.1001/jama.300.9.1027. PMID 18768414
- [Background] Barnes LL, Wilson RS, Li Y, Gilley DW, Bennett DA, Evans DA. Change in cognitive function in Alzheimer's disease in African-American and white persons. Neuroepidemiology. 2006;26(1):16-22. doi: 10.1159/000089231. Epub 2005 Oct 25. PMID 16254449
- [Background] Wilkins CH, Grant EA, Schmitt SE, McKeel DW, Morris JC. The neuropathology of Alzheimer disease in African American and white individuals. Arch Neurol. 2006 Jan;63(1):87-90. doi: 10.1001/archneur.63.1.87. PMID 16401740
- [Background] Larson EB, Wang L, Bowen JD, McCormick WC, Teri L, Crane P, Kukull W. Exercise is associated with reduced risk for incident dementia among persons 65 years of age and older. Ann Intern Med. 2006 Jan 17;144(2):73-81. doi: 10.7326/0003-4819-144-2-200601170-00004. PMID 16418406
- [Background] Kramer AF, Erickson KI, Colcombe SJ. Exercise, cognition, and the aging brain. J Appl Physiol (1985). 2006 Oct;101(4):1237-42. doi: 10.1152/japplphysiol.00500.2006. Epub 2006 Jun 15. PMID 16778001